CLINICAL TRIAL: NCT03484611
Title: Prediction of Metaphase II Oocytes According to Different Levels of Serum AMH in Poor Responders Using the Antagonist Protocol
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Maged, professor, Cairo University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 35
Record Dates: First submitted 2018-03-26; First posted 2018-04-02 (Actual); Last update posted 2018-04-02 (Actual); Status verified 2018-03

CONDITIONS: Invitro Fertilizaion
MeSH Terms: interventions — LHRH, Ac-Nal(1)-Cpa(2)-Trp(3)-Arg(6)-Ala(10)-; cetrorelix; Gonadotropins; Menotropins; Chorionic Gonadotropin; Embryo Transfer; Progesterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- AMH < 0.3 ng/ml (Active Comparator): Poor ovarian responders according to ESHRE consensus with serum AMH < 0,3 ng/ml
  Interventions: Drug: GnRH antagonist; Drug: Gonadotropins; Drug: Human chorionic gonadotropin; Procedure: Embryo transfer; Drug: Progesterone
- AMH 0.3 to 0.7 ng/ml (Active Comparator): Poor ovarian responders according to ESHRE consensus with serum AMH 0.3 to 0.7 ng/ml
  Interventions: Drug: GnRH antagonist; Drug: Gonadotropins; Drug: Human chorionic gonadotropin; Procedure: Embryo transfer; Drug: Progesterone
- AMH > 0.7 to 1 ng/ml (Active Comparator): Poor ovarian responders according to ESHRE consensus with serum AMH 0.7 to 1 ng/ml
  Interventions: Drug: GnRH antagonist; Drug: Gonadotropins; Drug: Human chorionic gonadotropin; Procedure: Embryo transfer; Drug: Progesterone

INTERVENTIONS:
Drug: GnRH antagonist — 0,25mg s.c, cetrotide, serono laboratories, Aubonne Switzerland) is given using flexible protocol, it is given when at least one follicle reaches size 14 mm to prevent premature lutenization ,until the day of hCG administration
  Other Names: cetrorelix
Drug: Gonadotropins — started on day 2 of the menstrual cycle until the day of HCG administration(choriomon,IBSA10000IU)with starting dose 300IU to 450IU
  Other Names: Human menopausal gonadotropin
Drug: Human chorionic gonadotropin — 10000 IU is given to induce final oocytes maturation when at least 2 follicles reached 14 mm or more
  Other Names: HCG
Procedure: Embryo transfer — 0ne to three grade 1 or 2 embryos were transferred on day 3 after oocyte retrieval. Embryo transfer was performed with a Wallace catheter (Smith Medical International Ltd, Hythe, Kent, UK)
Drug: Progesterone — vaginal prontogest 400 mg twice daily

SUMMARY:
A multicentric study looked into 179 poor responders who underwent antagonist protocol in ICSI cycles Gonadotrophines is started on day 2 with HMG until the day of HCG administration with starting dose 300IU to 450IU,with no pretreatment with OCPs or progestogens or estrogen.

GNRH antagonist (cetrorelix 0,25mg s.c, cetrotide, serono laboratories, Aubonne Switzerland) is given using flexible protocol, it is given when at least one follicle reaches size 14 mm to prevent premature lutenization ,until the day of hCG administration Ovarian ultrasound scans were performed using a 5.0-9.0 MHZ multi frequency trans vaginal probe to assess the ovarian response till the mature follicles reach18-20mm when hCG administration 10000 IU is given to induce final oocytes maturation , serum E2 is done on day of HCG trigger.

Trans vaginal ultrasound-guided oocyte retrieval is performed 34-36 hours after hCG injection.

Ultrasound -guided fresh embryo transfer is performed on day 3 or 5 after fertilization.

Progesterone support of luteal phase was commenced on the day of ovum pick up using prontogest 400 mg twice daily.

DETAILED DESCRIPTION:
A multicentric study looked into 179 poor responders who underwent antagonist protocol in ICSI cycles

Induction of ovulation cycle:

1. Gonadotrophines is started on day 2with HMG(merional, IBSA) ,until the day of HCG administration(choriomon,IBSA10000IU)with starting dose 300IU to 450IU,with no pretreatment with OCPs or progestogens or estrogen.
2. GNRH antagonist (cetrorelix 0,25mg s.c, cetrotide, serono laboratories, Aubonne Switzerland) is given using flexible protocol, it is given when at least one follicle reaches size 14 mm to prevent premature lutenization ,until the day of hCG administration
3. Ovarian ultrasound scans were performed using a 5.0-9.0 MHZ multi frequency trans vaginal probe (mindrayDP-5) to assess the ovarian response till the mature follicles reach18-20mm when hCG administration 10000 IU is given to induce final oocytes maturation , serum E2 is done on day of HCG trigger.
4. Trans vaginal ultrasound-guided oocyte retrieval is performed 34-36 hours after hCG injection.
5. Ultrasound -guided fresh embryo transfer is performed on day 3 or 5 after fertilization. . Embryo transfer was performed under abdominal ultrasound guide for proper embryo placement to the mid-uterine cavity. 0ne to three grade 1 or 2 embryos were transferred on day 3 after oocyte retrieval. The quality of the embryos were graded as 1,2,3 (1 being the best and 3 being the worst) based on the number of cells, degree of fragmentation and regularity. Embryo transfer was performed with a Wallace catheter (Smith Medical International Ltd, Hythe, Kent, UK). Progesterone support of luteal phase was commenced on the day of ovum pick up using prontogest 400 mg twice daily (IBSA, institut Biochemique,Switzerland).

ELIGIBILITY:
Inclusion Criteria:

* 3- On antagonist protocol 4- Poor responder according to ESHRE consensus; in which at least 2 of the following should be present:
* Advanced maternal age (≥ 40 years old) or any other risk factor
* A previous poor ovarian response (cycles cancelled or ≤ 3 oocytes with a conventional protocol)
* An abnormal ovarian reserve test (ORT); antral follicle count (AFC) < 5-7 follicles or anti-mullerian hormone (AMH) ≤0.5- 1.1 ng/ml NB: In the absence of advanced maternal age or abnormal ORT, two previous episodes of poor ovarian response after maximal stimulation patients are also considered poor responders according to ESHRE consensus.
* Presence and Adequate visualization of both ovaries
* Uterine cavity within normal anatomy

Exclusion Criteria:

Any factor which may affect reproductive outcome other than that the patient is a poor responder will be excluded from the study, like:

1. Severe male factor .
2. Uterine factor (eg: fibroid, polyp, Ashermann, .. etc)
3. Immunological disorder (eg: SLE, APS, … etc)
4. Thyroid or adrenal dysfunction
5. Neoplasia (especially: hypothalamic, pit, ovarian)
6. Women diagnosed with PCOS according to Rotterdam criteria
7. Hydrosalpinx that hasn't been surgically removed or ligated. 8 . Untreated hyperprolactinemia 9 . Abnormal bleeding disorder

10.Hepatic or renal dysfunction 11.Hypersenstivity to study medication ( GNRH antagonist) 12.Need to take medication that can influence ovarian stimulation 13.Endometriosis grade 3 or 4 14.Ovarian cyst> 10 cm.

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 179 (Estimated)
Dates: Start 2013-01 (Actual); Primary Completion 2018-04 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
Number of the retrieved oocytes | 34 hours after HCG injection
  number of oocytes retrieved 34 hours after HCG injection

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Maged, MD, Principal Investigator — professor
Locations (1):
- Kasr Alainy medical school, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided